CLINICAL TRIAL: NCT03602300
Title: A Phase 1, Open-Label, Four-Period, Two-Sequence, Two-Treatment, Single Dose, Randomized, Crossover Bioequivalence Study of a Test Tablet Formulation of Ravidasvir With the Reference Tablet Formulation of Ravidasvir in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: A Phase 1 Bioequivalence Study of a Test Tablet Formulation of Ravidasvir With the Reference Tablet Formulation of Ravidasvir Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-RDV-02-HCV
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Bioequivalence Study

STUDY DESIGN:
Intervention Model Description: A Phase 1, Open-Label, Four-Period, Two-Sequence, Two-Treatment, Single Dose, Randomized, Crossover Bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ravidasvir reference formulation (Active Comparator): Ravidasvir 200 mg oral single dose manufactured by EEPI
  Interventions: Drug: Ravidasvir reference formulation produced by EEPI
- Ravidasvir test formulation (Experimental): Ravidasvir 200 mg oral single dose manufactured by Doppel
  Interventions: Drug: Ravidasvir test formulation produced by Doppel

INTERVENTIONS:
Drug: Ravidasvir test formulation produced by Doppel — To compare the rate and extent of absorption for RDV when administered as a single 200 mg oral dose of the proposed commercial product ("test") produced by Doppel Farmaceutici with the clinical trial product ("reference") manufactured by EEPI in healthy volunteers, under fasted conditions.
  Arms: Ravidasvir test formulation
Drug: Ravidasvir reference formulation produced by EEPI — To compare the rate and extent of absorption for RDV when administered as a single 200 mg oral dose of the proposed commercial product ("test") produced by Doppel Farmaceutici with the clinical trial product ("reference") manufactured by EEPI in healthy volunteers, under fasted conditions.
  Arms: Ravidasvir reference formulation

SUMMARY:
In a phase 1, open-label, crossover study to evaluate the relative bioavailability of a tablet formulation of ravidasvir (test) versus the capsule formulation of ravidasvir (reference) in 24 healthy adult volunteers (PPI-668-104 study), relatively high intra-subject coefficients of variation were observed for both Cmax and AUC0-t.

A two-sequence, four-period replicate design will be used to allow the possibility to scale the acceptance range for Cmax if the observed intra-subject coefficient of variation for the reference formulation is greater than 30%

DETAILED DESCRIPTION:
During the course of development, a new batch of ravidasvir tablets has been prepared by the proposed commercial manufacturer (Doppel Farmaceutici, Italy). Tablets manufactured by Doppel Farmaceutici are intended to be used in subsequent clinical trials and be registered as the commercial product. The purpose of this Phase 1, Open-Label, Four-Period, Two-Sequence, Two-Treatment, Single Dose, Randomized, Crossover Bioequivalence Study is to assess if ravidasvir 200 mg tablets supplied by European Egyptian Pharmaceutical Industries (EEPI) and tablets from Doppel Farmaceutici are bioequivalent.

Primary objectives:

To compare the rate and extent of absorption for ravidasvir (RDV) when administered as a single 200 mg oral dose of the proposed commercial product ("test") produced by Doppel Farmaceutici with the clinical trial product ("reference") manufactured by EEPI in healthy volunteers, under fasted conditions.

Secondary objectives To evaluate the safety and tolerability of single oral doses of RDV in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Must be between 18 and 55 years of age, inclusive.
* Must be a non-smoker. The use of nicotine or nicotine-containing products must be discontinued 90 days prior to the first dose of study drug. Users of electronic cigarette are not allowed to participate in this study. A smokerlyzer test will be performed to estimate the amount of carbon monoxide in the breath.
* Must have a calculated body mass index (BMI) of 18.0 to 29.9 kg/m2.
* Must be HIV-1 antibody negative.
* Must be hepatitis B (HBV) surface antigen negative.
* Must be hepatitis C (HCV) antibody negative.
* Females of childbearing potential must have a negative serum pregnancy test at Screening and on Day 0.
* Females of childbearing potential must agree to utilize highly effective contraception methods (with the exception of hormonal contraceptive) from 3 weeks prior to baseline (Day 0) throughout the duration of study treatment and for 30 days following the last dose of study drug. Female healthy volunteers who utilize hormonal contraceptive as one of their birth control methods are not allowed to participate in this study.
* Men who participate in this study must not father a child and must agree to use contraceptive protection in the form of a double barrier method (condom or diaphragm) from the moment they sign the ICF until the Post-Study Safety Assessment.
* Healthy volunteers must, in the opinion of the Investigator, be in good health based upon medical history, physical examination (including vital signs), and screening laboratory evaluations (haematology, chemistry, and urinalysis) must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance.
* Have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the Investigator.
* Must have negative urine screen for drugs of abuse (including ketamine, amphetamines, tetrahydrocannabinol, morphine, methamphetamine, and benzodiazepines)
* Must be willing and able to comply with all study requirements

Exclusion Criteria:

* Healthy volunteers with any hematologic or urinary analyte that is outside the normal limits of the study laboratory and have been determined by the Investigator to have clinical significance at Screening will be excluded
* Pregnant or lactating female healthy volunteers.
* Have any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include renal, cardiac, hematologic, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central or peripheral nervous, gastrointestinal (including an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), or immunodeficiency disorders, active infection, or malignancy that is clinically significant or requiring treatment.
* Have participated in an investigational trial involving administration of any investigational compound within 90 days prior to the study dosing or 5-times the half-life of the drug tested in the previous clinical trial, whichever is longer (time calculated relative to the last dose in the previous clinical trial).
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance.
* Have poor venous access and unable to donate blood.
* Have donated or lost blood (≥500ml) within two months of study dosing.
* Have donated plasma within 7 days of study dosing.
* Have difficulty in swallowing solids like tablets.
* Have taken any prescription medications or over-the-counter medications including herbal products within 1 week of commencing study drug dosing with the exception of vitamins and/or acetaminophen and/or ibuprofen.
* Female healthy volunteers who utilize hormonal contraceptive as one of their birth control methods.
* Have a history of significant drug allergy.
* Smokers and users of electronic cigarette.
* Unable to comply with study requirements.
* Believed by the study Investigator to be inappropriate for study participation for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
RDV Plasma CMax when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  Plasma RDV Cmax will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose
RDV area under the plasma concentration-time curve from time of intake until infinity (AUC0-∞) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  Area under the plasma concentration-time curve from time of intake until infinity (AUC0-∞) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV area under the plasma concentration-time curve from time of intake until the last quantifiable concentration (AUC0-t) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  Area under the plasma concentration-time curve from time of intake until the last quantifiable concentration (AUC0-t) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.

SECONDARY OUTCOMES:
RDV maximum plasma concentration (tmax) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV maximum plasma concentration (tmax) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV mean residence time (MRT) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV mean residence time (MRT) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV elimination rate constant (λz) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV elimination rate constant (λz) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV elimination half-life (t1/2, estimated based on λz), when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV elimination half-life (t1/2, estimated based on λz) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV apparent volume of distribution when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV apparent volume of distribution will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV terminal phase (Vz/F) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV terminal phase (Vz/F) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV apparent clearance (CL/F) when administered as a single 200 mg oral dose of the test versus reference product | Measurement within 48 hours post-dose
  RDV apparent clearance (CL/F) will be calculated based on plasma RDV concentrations at pre-dose (time 0 hours) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, and 48 hours post-dose.
RDV safety (Incidence of treatment-related adverse events as assessed by CTCAE v4.03) when administered as a single 200 mg oral dose of the test versus reference product | From 1st patient consent until last patient completes the post-study safety assessment over a total period of 60 days
  Safety will be assessed by monitoring clinical adverse events (AEs) incidence
RDV tolerability (Incidence of treatment-related adverse events as assessed by CTCAE v4.03) when administered as a single 200 mg oral dose of the test versus reference product | From 1st patient consent until last patient completes the post-study safety assessment over a total period of 60 days
  Tolerability will be assessed by monitoring clinical adverse events (AEs) incidence

CONTACTS AND LOCATIONS:
Overall Officials: Damenthi Nair, MD, Principal Investigator — KPJ Ampang Puteri Specialist Hospital
Locations (1):
- Ampang hospital, Ampang, Selangor, Malaysia